CLINICAL TRIAL: NCT01498965
Title: BASELINE: Babies After Scope: Evaluating the Longitudinal Impact Using Neurological and Nutritional Endpoints
Brief Title: The Cork BASELINE Birth Cohort Study
Acronym: BASELINE
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: National Children's Research Centre, Ireland (Network)
Collaborators: Food Standards Agency, United Kingdom (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2185
Record Dates: First submitted 2011-12-20; First posted 2011-12-26 (Estimated); Last update posted 2015-01-21 (Estimated); Status verified 2015-01

CONDITIONS: Food Allergy; Eczema; Obesity
Keywords: food allergy; eczema; Vitamin D status; body composition; obesity; neurodevelopmental and behavioural outcome
MeSH Terms: conditions — Food Hypersensitivity; Eczema; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — MAternal DNA, plasma, serum and urine Umbilical serum, plasma, DNA, RNA At 2 years and 5 years: serum, and DNA
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The Departments of Paediatrics and Child Health, Obstetrics/Gynaecology and Nutritional Sciences, University College Cork, and the Department of Dermatology, Trinity College, Dublin have a unique and urgent opportunity to form a birth cohort of over 2000 children whose growth and maternal health status will have been closely monitored from early pregnancy. Longitudinal monitoring of these infants will allow direct investigation of several research areas in a way which has not previously been possible in Ireland, or abroad. The investigators propose to focus on three main research themes: the effects of intrauterine growth restriction, the incidence and prevalence of food allergy and eczema in early childhood and the incidence and effects of maternal and infant vitamin D status on the growth and health of Irish children. Although the investigators initial proposal will focus on these important areas, the formation of this birth cohort will offer many opportunities for further research as the cohort grows older. It will form a unique bio-bank of information from Irish children collected longitudinally from soon after their conception. The mothers of these infants are currently being recruited, which leaves us with a narrow window of opportunity to put in place a pathway of investigation for these children. To ignore this opportunity would be to lose access to a wealth of information regarding child health and disease. The potential for this cohort to provide definitive answers to current, and future, theories of disease causation is enormous.

DETAILED DESCRIPTION:
SPECIFIC AIMS:

Our underlying aim is to establish a prospective paediatric birth cohort which will have access to detailed information on maternal health, fetal growth, and childhood nutrition, growth and development in the first 2 years of life. This cohort will have the advantage of a stored biobank of maternal and fetal plasma, serum and DNA. This cohort will allow us to monitor the effects of intrauterine growth and nutrition on early life illnesses.

Our specific aims are:

1. To establish the fetal and early life growth trajectories which foretell later neurocognitive disability and metabolic disorder
2. To establish the incidence and prevalence of food allergy and eczema in Irish children and investigate the relationship between Vitamin D deficiency and allergic disorders of early childhood.
3. To establish the prevalence of maternal and neonatal vitamin D deficiency in an Irish paediatric population

Introduction:

There is increasing evidence that the intrauterine environment has important effects, not only on fetal growth, but also on the life-long health of the child. A term infant is the end result of nine months of immunological and nutritional interplay between the fetus, placenta and mother. Therefore, it is not surprising that this nutritional and hormonal environment has far-reaching effects on childhood health and adult health risk. Fetal nutritional status has been repeatedly linked with adult risk of hypertension, hypercholesterolaemia, Type 2 diabetes and cardiovascular disease. Fetal growth restriction may be associated with neurocognitive delay and long term behavioural problems. We know that maternal vitamin D status has a direct effect on bone growth, not just in neonates, but also on the bone mass and fracture risk of the adolescent offspring. More recently there is some evidence that maternal vitamin D and E deficiency may contribute to a substantial proportion of the increasing incidence of childhood asthma. It is clear, then, that to establish the pathophysiology of many childhood diseases we will need to look back to long before birth.

Previous large birth cohorts in the UK have added greatly to our current knowledge of paediatric health and disease. However the early ALSPAC cohort study examining the "Children of the Nineties" did not have access to the detailed and serial fetal scanning which the SCOPE study will provide to BASELINE. The more recent Southampton Women's Study recruited a similar number of maternal and fetal dyads. The SWS study protocol included fetal scanning and stored DNA, but does not have a cord biobank of serum and plasma samples. The BASELINE study will have access to maternal blood sampling, detailed health questionnaires, serial fetal scanning and multiple aliquots of stored umbilical cord blood. In addition our study will provide reference data in Irish children, something which overseas cohorts can not provide to Irish health care planners and providers.

We believe that the BASELINE study is Ireland's opportunity to establish a longitudinal birth cohort with the potential to answer important questions in the study of diseases in early life, later childhood and beyond. We will be able to identify risk factors for common disorders such as diabetes, eczema and asthma. The BASELINE genetic biobank will allow us to examine candidate genetic markers of disorders as they arise in the cohort. This study has the potential to transform the landscape of paediatric research in Ireland.

ELIGIBILITY:
Inclusion Criteria:

* All liveborn infants whose mothers were recruited to the SCOPE Ireland study at 15 weeks gestation.
* Singleton pregnancies, no previous history or risk of pre-eclampsia

Exclusion Criteria:

* Stillbirths, or mothers who do not consent to paediatric follow up.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All infants born to mothers enrolled in the SCOPE pregnancy study (www.scopestudy.net) in SCOPE Ireland. First time, low risk mothers with singleton pregnancies.
Sampling Method: Probability Sample
Enrollment: 2185 (Actual)
Dates: Start 2008-08; Primary Completion 2016-10 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
To establish a longitudinal birth cohort study to examine early life environment and effect on childhood illness | 24 months

SECONDARY OUTCOMES:
To establish the prevalence of maternal and neonatal vitamin D deficiency in an Irish paediatric population | 24 months
  Maternal vitamin, Vitamin D at birth in umbilical cord blood, and at 24 months of age
To establish the incidence and prevalence of food allergy and eczema in Irish children and investigate the relationship between Vitamin D deficiency and allergic disorders of early childhood | 24 months
  To establish the early life factors, including parental allergy, genetic susceptibility measured using Fillagrin mutational status,skin barrier function and vitamin D status and their effect on risk of eczema and food allergy in the first 2 years of life.
To establish the fetal and early life growth trajectories which foretell later neurocognitive disability and metabolic disorder | 24 months
  To examine the relationship between in-utero growth, measured using body composition, and customised birth weight centiles and nerudevelopmental outcome at 24 months. We will also examin risk factors for childhood obesity and metabolic dysfunction at 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Deirdre M Murray, MD. PhD, Principal Investigator — University College Cork; Jonathan OB Hourihane, MD, Study Director — University College Cork; Louise K Kenny, PhD, Study Director — University College Cork; Mairead Kiely, PhD, Study Director — University College Cork; Alan Irvine, MD. PhD, Study Director — University of Dublin, Trinity College
Locations (1):
- Department of Paediatrics and Child Health, Cork University Hospital, Cork, Ireland

REFERENCES:
- [Result] Hawkes CP, Hourihane JO, Kenny LC, Irvine AD, Kiely M, Murray DM. Gender- and gestational age-specific body fat percentage at birth. Pediatrics. 2011 Sep;128(3):e645-51. doi: 10.1542/peds.2010-3856. Epub 2011 Aug 8. PMID 21824882
- [Result] O'Donovan SM, Murray DM, Hourihane JO, Kenny LC, Irvine AD, Kiely M. Cohort profile: The Cork BASELINE Birth Cohort Study: Babies after SCOPE: Evaluating the Longitudinal Impact on Neurological and Nutritional Endpoints. Int J Epidemiol. 2015 Jun;44(3):764-75. doi: 10.1093/ije/dyu157. Epub 2014 Aug 7. PMID 25102856
- [Result] Kelleher MM, O'Carroll M, Gallagher A, Murray DM, Dunn Galvin A, Irvine AD, Hourihane JO. Newborn transepidermal water loss values: a reference dataset. Pediatr Dermatol. 2013 Nov-Dec;30(6):712-6. doi: 10.1111/pde.12106. Epub 2013 Mar 5. PMID 23458265
- [Derived] O'Connor C, Livingstone V, O'B Hourihane J, Irvine AD, Boylan G, Murray D. Early emollient bathing is associated with subsequent atopic dermatitis in an unselected birth cohort study. Pediatr Allergy Immunol. 2023 Jul;34(7):e13998. doi: 10.1111/pai.13998. PMID 37492907
- [Derived] McCarthy EK, Murray DM, Malvisi L, Kenny LC, O'B Hourihane J, Irvine AD, Kiely ME. Antenatal Vitamin D Status Is Not Associated with Standard Neurodevelopmental Assessments at Age 5 Years in a Well-Characterized Prospective Maternal-Infant Cohort. J Nutr. 2018 Oct 1;148(10):1580-1586. doi: 10.1093/jn/nxy150. PMID 30169669
- [Derived] Norris T, McCarthy FP, Khashan AS, Murray DM, Kiely M, Hourihane JO, Baker PN, Kenny LC; SCOPE Ireland Cohort study and the Cork BASELINE Birth Cohort Study. Do changing levels of maternal exercise during pregnancy affect neonatal adiposity? Secondary analysis of the babies after SCOPE: evaluating the longitudinal impact using neurological and nutritional endpoints (BASELINE) birth cohort (Cork, Ireland). BMJ Open. 2017 Dec 1;7(11):e017987. doi: 10.1136/bmjopen-2017-017987. PMID 29196482
- [Derived] Denihan NM, Looney A, Boylan GB, Walsh BH, Murray DM. Normative levels of Interleukin 16 in umbilical cord blood. Clin Biochem. 2013 Dec;46(18):1857-9. doi: 10.1016/j.clinbiochem.2013.07.012. Epub 2013 Jul 24. PMID 23891891
- [Derived] Walsh BH, Boylan GB, Livingstone V, Kenny LC, Dempsey EM, Murray DM. Cord blood proteins and multichannel-electroencephalography in hypoxic-ischemic encephalopathy. Pediatr Crit Care Med. 2013 Jul;14(6):621-30. doi: 10.1097/PCC.0b013e318291793f. PMID 23823198
- [Derived] Walsh BH, Broadhurst DI, Mandal R, Wishart DS, Boylan GB, Kenny LC, Murray DM. The metabolomic profile of umbilical cord blood in neonatal hypoxic ischaemic encephalopathy. PLoS One. 2012;7(12):e50520. doi: 10.1371/journal.pone.0050520. Epub 2012 Dec 5. PMID 23227182
- See also: The Cork BASELINE Birth Cohort Study home page — http://www.baselinestudy.net
- See also: SCOPE pregnancy study — http://www.scopestudy.net